CLINICAL TRIAL: NCT02549677
Title: Comparison the Safety and Efficacy of Epirubicin Plus Cyclophosphamide (EC)Versus Docetaxel Plus Cyclophosphamide (TC) in Lymph Node Negative, ER Positive, Her2 Negative Breast Cancer Patients as Adjuvant Chemotherapy
Brief Title: Epirubicin Versus Docetaxel Plus Cyclophosphamide in Lymph Node Negative, ER-positive, Her2-negative Breast Cancer
Acronym: ELEGANT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Li Zhu, doctor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJBC1506
Record Dates: First submitted 2015-09-06; First posted 2015-09-15 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Anthracyclines; Docetaxel; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EC regimen (Experimental): Epirubicin, cyclophosphamide
  Interventions: Drug: Epirubicin; Drug: cyclophosphamide
- TC regimen (Active Comparator): docetaxel, cyclophosphamide
  Interventions: Drug: Docetaxel; Drug: cyclophosphamide

INTERVENTIONS:
Drug: Epirubicin — epirubicin, 90mg per square meter, every 3 weeks, day 1
  Other Names: anthracycline
  Arms: EC regimen
Drug: Docetaxel — docetaxel, 75mg per square meter, every 3 weeks, day 1
  Other Names: taxotere
  Arms: TC regimen
Drug: cyclophosphamide — cyclophosphamide, 600mg per square meter, every 3 weeks, day 1

SUMMARY:
The purpose of this study is to compare the safety and efficacy of epirubicin plus cyclophosphamide versus docetaxel plus cyclophosphamide in lymph node negative, estrogen receptor (ER) positive, human epithelial growth factor receptor 2 (HER2) negative breast cancer patients as adjuvant chemotherapy.

DETAILED DESCRIPTION:
This is a non-inferiority study. According to previous study results, the investigators hypothesize the incidence of grade 3-4 neutropenia is 40%, with a α of 0.05 and β of 0.8, a sample size of 264 cases if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥18 years and < 70 years with life expectancy > 12 months
2. Have finished radical operation, pathologically verified no lymph node involvement
3. Operation specimens are available for ER, progesterone receptor (PR) and Her2 detection, patients should be with ER positive, Her2 negative tumor.
4. Adequate bone marrow function
5. Adequate liver and renal function
6. Has Eastern Cooperative Oncology Group (ECOG0 Performance Score 0-1;
7. Women with potential child-bearing must have a negative pregnancy test (urine or serum) within 7 days of drug administration and agree to use an acceptable method of birth control to avoid pregnancy for the duration of the study;
8. Written informed consent according to the local ethics committee requirements.

Exclusion Criteria:

1. Prior systemic or loco-regional treatment of breast cancer, including chemotherapy;
2. Metastatic breast cancer;
3. With a history of malignant tumor except uterine cervix cancer in situ or skin basal cell carcinoma;
4. Patients with medical conditions that indicate intolerant to adjuvant chemotherapy and related treatment, including uncontrolled pulmonary disease, diabetes mellitus, severe infection, active peptic ulcer, coagulation disorder, connective tissue disease or myelo-suppressive disease;
5. Has active hepatitis B or hepatitis C with abnormal liver function tests (LFTs) or is known to be HIV positive;
6. History of congestive heart failure, uncontrolled or symptomatic angina pectoris, arrhythmia or myocardial infarction; poorly controlled hypertension;
7. Has peripheral neuropathy ≥ grade 1;
8. Patient is pregnant or breast feeding;
9. Known severe hypersensitivity to any drugs in this study;
10. Treatment with any investigational drugs within 30 days before the beginning of study treatment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2015-10; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
number of participants with grade 3-4 neutropenia assessed by CTCAE v4.0 | up to 16 weeks
  number of participants with neutrophil count less than 1000 per milliliter

SECONDARY OUTCOMES:
number of participants with grade 3-4 leukopenia assessed by CTCAE v4.0 | up to 16 weeks
  number of participants with leukocyte count less than 2000 per milliliter
number of participants with febrile neutropenia assessed by CTCAE v4.0 | up to 16 weeks
  number of participants with neutropenia count less than 1000 per milliliter and temperature highe than 38.5℃
breast cancer relapse | three years
  number of participants with any locoregional recurrence, contralateral breast cancer or distant metastasis
all cause mortality | three years
  number of participans died from all cause

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhu, doctor, Principal Investigator — Shanghai Jiao Tong University School of Medicine affiliated Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD